CLINICAL TRIAL: NCT05203354
Title: Omentin-1 Level in Psoriatic Patients Treated With Narrowband Ultraviolet B Phototherapy Versus Acitretin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahmoud Ahmed Ali Ahmed (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Ahmed Ali Ahmed, Assistant lecturer, Aswan University Hospital
Organization: Aswan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 288/9/18
Record Dates: First submitted 2021-12-14; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Acitretin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- NB-UVB group (Active Comparator): Patients who receive Narrowband ultraviolet B phototherapy
  Interventions: Radiation: Narrowband Ultraviolet B
- Acitretin group (Active Comparator): Patients who receive acitretin
  Interventions: Drug: Acitretin
- Control group (No Intervention): It includes apparently healthy people who will be compared to patients in the measurement of Omentin-1 level

INTERVENTIONS:
Radiation: Narrowband Ultraviolet B — patients will exposed to sessions of NB-UVB phototherapy twice weekly for 3 months
  Other Names: NB-UVB phototherapy
  Arms: NB-UVB group
Drug: Acitretin — patients will received acitretin in dose 0.5-1 mg/kg daily for 3 months
  Arms: Acitretin group

SUMMARY:
Studying the effects of Narrowband Ultraviolet B versus acitretin on psoriatic patients

DETAILED DESCRIPTION:
Compare the effects of Narrowband Ultraviolet B versus acitretin on serum Omentin-1 level in psoriatic patients as case control study by dividing patients into 3 groups: group 1 include patients receive Narrowband Ultraviolet B, group II includes patients receive acitretin (0.5-1 mg/day) and control group. The duration of this study about 3 months after receving those interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes with psoriasis vulgaris.

Exclusion Criteria:

* • Patients with history of malignancies, renal and liver diseases.

  * Patients received NB-UVB phototherapy in the last 6 months.
  * Patients treated with methotrexate or biologic agents and any systemic treatment of psoriasis.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Decrease Omentin-1 serum level in both groups treated with NB-UVB and Acitretin | 3 months
  This outcome indicates potential role of Omentin-1 in psoriasis pathogenesis and its involvement in pathogenesis of obesity and related diseases as metabolic syndrome. So it will be concluded that high levels of this protein could be marker against obesity and related disorders including psoriasis. Omentin-1 can be valuable marker for psoriasis severity detected by its correlation with psoriasis area severity index (PASI) score and for evaluating the therapeutic outcomes

SECONDARY OUTCOMES:
Decrease PASI score in psoriatic patients | 3 months
  Decrease in PASI score in psoriatic patients after treatment with NB-UVB acitretin

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine - Aswan university, Aswān, Egypt